CLINICAL TRIAL: NCT02346318
Title: The Randomized Controlled Clinical Trial of Kushen Injection Reducing Radiotherapy Related Adverse Reactions in Lung Cancer
Brief Title: The Randomized Controlled Clinical Trial of Kushen Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Zheng Ju Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014EC085-01
Record Dates: First submitted 2014-12-04; First posted 2015-01-27 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2014-10

CONDITIONS: Lung Cancer
Keywords: Radiotherapy; Adverse Effect; Dermatitis or Eczema
MeSH Terms: conditions — Lung Neoplasms; Dermatitis; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KS injection arm (Experimental): Radiation and chemotherapy and compound Kushen Injection
  Interventions: Drug: Compound Kushen Injection
- Control arm (No Intervention): Radiation and chemotherapy

INTERVENTIONS:
Drug: Compound Kushen Injection — Compound Kushen Injection 20ml i.v.drip qd, synchronize with radiotherapy, total dosage is 400ml.
  Other Names: KS injection
  Arms: KS injection arm

SUMMARY:
The randomized controlled multicenter clinical study of compound Kushen Injection to reduce the radiotherapy related adverse reactions in lung cancer is a phase Ⅳ clinical trials，The main purpose is to evaluate the effect of compound Kushen Injection in preventing and reducing the radiotherapy related adverse reactions. The participants of the clinical trials are patients with lung cancer who need thoracic radiotherapy. In clinical trials, one group of participants is given compound Kushen Injection with chemoradiotherapy, while another group is only given chemoradiotherapy. The period of trials is 18 months.

DETAILED DESCRIPTION:
Patients with lung cancer who need thoracic radiotherapy will be enrolled in the trial, then seprated randomly in two group,the KS injection group treated with chemoradiotherapy plus KS injection; the contral group treated with chemoradiotherapy only. After 6 months observation, The rates of incidence and the degree of adverse reactions caused by redioterapy; the completion rate of radiotherapy; clinical Symptoms; Qof and pulmonary function tests etc. will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Before the start of the study, All patients have been fully understood the reseach and the must sign the informed consent
* To be aged from 18 to 75 years old, both gender
* The lung cancer diagnosis must be proved by pathology
* According to RECIST (version 1.1), At least 1 objectively measurable Tumor lesion (iconography: CT, MRI), the assessable lesion can be measured accurately, maximum diameter more than at least 10mm (Malignant lymph nodes on CT scans short diameter less than at least 15 mm)
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Lung function FEV1 more than at least 1Land more than 50% A normal value
* The function of each organ is basically normal :ANC more than 1.5*10^9/L, Platelet count more than 100*10^9/L, Hb more than 9.0g/dl, BIL at normal level or less than 1.5*ULN, AST (SGOT), ALT (SGPT) less than 2.5*ULN(less than 5*ULN, if with liver metastases), SCr less than 1.5*ULN
* The expected survival tme must more than 6 months.

Exclusion Criteria:

* Lung or mediastinal have received radiotherapy before or ever treated with Compound Kushen Injection within 2weeks
* Pregnancy or lactation women
* Patients with severe, uncontrolled organic lesions or infection, such as decompensated heart, lung, kidney failure can lead to tolerance of chemotherapy - Participating or within the last 30 days participated in other clinical trials
* Hypersensitiveness to any kind of trial regime
* Had a history of serious Psychological or Psychiatric disorders, Drug addiction or Alcohol dependence
* Estimating the compliance of patients to participate in this clinical trial is insufficient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The rates of incidence and the degree of adverse reactions caused by redioterapy | 6 months
  radio-pulmonary lesion,radiation esophagitis,Radiation Induced Heart Disease

SECONDARY OUTCOMES:
The completion rate of radiotherapy | 2 months
  Compare two groups of patients with completion of the radiotherapy plans
Clinical Symptoms (MDASI-TCM) | 6 months
  MDASI-TCM
Quality of Life (EORTC QLQ-C30) | 6 months
  EORTC QLQ-C30
ECOG PS (ECOG PS score) | 6 months
  ECOG PS score
Weight | 6 months
  After the treatment,Healing after weight 1 kg to "add",Reduce 1 kg to "fall",Less than 1 kg of change as a "stable"
Gene molecule detection (EGFR) | 4 weeks
  EGFR
Pulmonary function tests (FEV1,FVC,DLCO) | 6 months
  FEV1,FVC,DLCO
Immune function (Observation indexes including NK、T lymphocyte subpopulation（CD3、CD4、CD8）、CD4/CD8) | 6 months
  Observation indexes including NK、T lymphocyte subpopulation（CD3、CD4、CD8）、CD4/CD8

CONTACTS AND LOCATIONS:
Overall Officials: Shuanghu Yuan, postdoctoral, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong cancer hospital, Jinan, Shandong, China